CLINICAL TRIAL: NCT03037645
Title: A Phase 1b/2 Dose-Escalation and Cohort-Expansion Study of the Noncovalent, Reversible Bruton's Tyrosine Kinase Inhibitor, SNS-062, in Patients With B-Lymphoid Malignancies
Brief Title: Safety, PK, PD, and Antitumor Activity of Vecabrutinib (SNS-062) in B Lymphoid Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Phase 1b portion completed. Sponsor decided not to proceed with P2 portion of study. Vecabrutinib was very well tolerated, there was insufficient evidence of activity at the doses tested in the Phase 1b to advance to Phase 2.
Sponsor: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 062-HEM-102
Record Dates: First submitted 2017-01-25; First posted 2017-01-31 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Lymphoplasmacytoid Lymphoma; Mantle-Cell Lymphoma; Waldenstrom Macroglobulinemia; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma
Keywords: CLL; hematological diseases; relapsed; cancer; malignancy; SNS-062; B-lymphoid; chronic lymphocytic leukemia; small lymphocytic lymphoma; lymphoplasmacytoid lymphoma; Waldenström's macrogloulinemia; mantle cell lymphoma; SLL; LPL; WM; MCL; refractory; DLBCL-ABC; DLBCL; follicular lymphoma; diffuse large B-cell lymphoma; CLL/SLL; MZL; marginal zone lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Hematologic Diseases; Recurrence; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalating cohorts of SNS-062 (Experimental): Sequential groups, 25, 50, 100, 200, 300, 400 and 500 mg twice daily to determine maximum tolerated dose and recommended dose (RD) in the treatment of various hematological cancers followed by expansion of the recommended dose cohort in Phase 2 of the study treating hematological cancers.
  Interventions: Drug: SNS-062

INTERVENTIONS:
Drug: SNS-062 — SNS-062 will be orally administered twice daily and available in capsules containing either 25 mg or 100 mg of active ingredient.

SUMMARY:
This is an open-label Phase 1b/2 study in patients with chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL)or non hodgkin's lymphoma (NHL) who have failed prior standard of care therapies including a BTK inhibitor where one is approved for the indication.

DETAILED DESCRIPTION:
This study includes 2 parts: phase 1 (dose escalation) and phase 2 (cohort expansion) in patients with CLL/SLL or NHL who have failed prior standard of care therapies including a BTK inhibitor where one is approved for the indication. NHL indications include lymphoplasmacytoid lymphoma/Waldenström's macroglobulinemia (LPL/WM), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), diffuse large B-cell lymphoma of the activated B-cell subtype (DLBCL-ABC), and follicular lymphoma (FL). In Phase 1b, cohorts of 3 to 6 patients are studied at each dose level, starting with 25 mg vecabrutnib BID in oral capsule form. Following identification of the MTD and/or recommended dose, in Phase 2 only CLL/SLL patients will be enrolled to expansion cohorts to further characterize the clinical activity, safety, and pharmacology of vecabrutinib. Cycle length is 4 weeks.

ELIGIBILITY:
Inclusion Criteria (Key factors listed):

* Eastern Cooperative Oncology Group Performance Status of ≤2.
* Confirmed malignancy with relapsed/refractory disease after ≥2 lines of standard systemic therapy including prior BTK inhibitor therapy having CLL, LPL/WM, MCL or MZL and for DLBCL-ABC and FL, after ≥2 lines of standard systemic therapy (Phase 1b). For Phase 2, CLL/SLL patients with confirmed malignancy with relapsed/refractory disease after ≥1 line of standard systemic therapy including prior BTK inhibitor therapy
* Presence of measurable disease through various assessments depending on specific cancer type.
* Current medical need for therapy of the B-lymphoid malignancy.

Exclusion Criteria (Key factors listed):

* Active central nervous system involvement.
* History of second primary malignancy that has progressed or required systemic treatment in the past 2 years. Exceptions include: local cancers of the skin, cervix or breast cancers, non-invasive bladder cancer, hormone sensitive prostate cancer with stable PSA ≥3 months, and other localized solid tumors in situ/other low risk cancers.
* Significant cardiovascular disease or electrocardiogram (ECG) abnormalities
* Ongoing risk for bleeding due to bleeding diathesis, platelet function disorder, uncontrolled peptic ulcer disease, oral anticoagulation medications.
* Evidence of uncontrolled systemic bacterial, fungal or viral infections at the start of drug therapy.
* Demonstrated intolerance to BTK inhibitor as shown by discontinuation due to adverse effects.
* Use of a moderate or strong inhibitor or inducer of CYP3A4 within 7 days prior to start of study therapy (e.g., some antibiotics, antifungals, anticonvulsants, grapefruit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and/or Recommended dose of SNS-062 (Phase 1b) | Up to approximately 21 months
  To determine the Maximum Tolerated Dose (MTD) and/or Recommended Dose (RD)within the tested SNS-062 dose range. The MTD is the highest tested dose level at which ≥6 subjects have been treated and which is associated with a Cycle 1 dose limiting toxicity (DLT) in <33% of the subjects. The RD may be the MTD or may be a lower dose.
Objective Response Rate (ORR) (Phase 2) | Up to approximately 36 months
  Phase 2 portion of study measuring ORR and corresponding 90% confidence intervals by cohort. ORR will be defined by disease subtype as the proportion of subjects who achieve CLL/SLL: a CR, CRi, or PR.

SECONDARY OUTCOMES:
Safety as assessed through reported AEs, SAEs, DLTs and abnormal lab findings (Phase 1b and Phase 2) | Up to approximately 36 months
  Type, severity, timing of onset, duration, and relationship to study drug of any TEAEs or abnormalities of laboratory tests, SAEs, DLTs, or AEs leading to study discontinuation.
Characterization of Pharmacokinetics (AUC) (Phase 1b and Phase 2) | Up to approximately 36 months
  Area Under the Curve (AUC)
Characterization of Pharmacokinetics (Cmin,ss) (Phase 1b and Phase 2) | Up to approximately 36 months
  Minimum Plasma Concentration During Dosing Interval at Steady-State (Cmin,ss)
Characterization of Pharmacokinetics (Cmax) (Phase 1b and Phase 2) | Up to approximately 36 months
  Maximum Plasma Concentration (Cmax)
Characterization of Pharmacokinetics (Tmax) (Phase 1b and Phase 2) | Up to approximately 36 months
  Time of Maximum Plasma Concentration (Tmax)
Preliminary evidence of anti-tumor activity, in terms of Time to Response (TTR) as assessed by the Investigator. (Phase 2) | Up to approximately 36 months
  Measure of Time to Response (TTR) as evaluated by standard response and progression criteria for CLL/SLL.
Preliminary evidence of anti-tumor activity, in terms of Duration of Response (DOR) as assessed by the Investigator. (Phase 2) | Up to approximately 36 months
  Measure of Duration of Response (DOR) as evaluated by standard response and progression criteria for CLL/SLL.
Preliminary evidence of anti-tumor activity, in terms of Response Rate (RR) as assessed by the Investigator. (Phase 2) | Up to approximately 36 months
  Measure of Response Rate (RR) as evaluated by standard response and progression criteria for CLL/SLL.
Preliminary evidence of anti-tumor activity, in terms of Disease Control Rate (DCR) as assessed by the Investigator. (Phase 2) | Up to approximately 36 months
  Measure of Disease Control Rate (DCR) as evaluated by standard response and progression criteria for CLL/SLL.
Preliminary evidence of anti-tumor activity, in terms of Progression-Free Survival (PFS) as assessed by the Investigator. (Phase 2) | Up to approximately 36 months
  Measure of Progression-Free Survival (PFS) as evaluated by standard response and progression criteria for CLL/SLL.
Preliminary evidence of anti-tumor activity, in terms of Overall Survival (OS) as assessed by the Investigator. (Phase 2) | Up to approximately 36 months
  Measure of Overall Survival (OS) as evaluated by standard response and progression criteria for CLL/SLL.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Acton, MD, Study Director — Sunesis Pharmaceuticals
Locations (11):
- United States (11):
  - University of California Irvine Medical Center, Orange, California
  - UC San Diego Moores Cancer Center, San Diego, California
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medicine, New York, New York
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557